CLINICAL TRIAL: NCT00183300
Title: Effectiveness of Prolonged Exposure Therapy on Reducing Neuroendocrine-Related Symptoms of Post-Traumatic Stress Disorder in Women
Brief Title: Relationship Between the Biological and Psychological Correlates of PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH062003 (NIH); R01MH062003 (NIH); DATR AD-TS
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2007-12

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post-traumatic stress disorder; PTSD; Prolonged Exposure; Cognitive-Behavior Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy

SUMMARY:
This study will determine the effectiveness of immediate treatment with prolonged exposure therapy (PE) versus delaying treatment with PE in altering neuroendocrine-related symptoms of post-traumatic stress disorder in women.

DETAILED DESCRIPTION:
Post-Traumatic Stress Disorder (PTSD) is a psychiatric disorder that can occur following exposure to a traumatic incident in which grave physical harm occurred or was threatened. PTSD is marked by clear biological changes as well as psychological symptoms. Many people with PTSD repeatedly relive the trauma in the form of flashback episodes, memories, nightmares, or frightening thoughts. Chronic PTSD can also affect the neuroendocrine system by altering functionality of some chemicals in the brain, including cortisol and catecholamines (e.g., norepinephrine). This study will determine the effectiveness of immediate treatment with prolonged exposure therapy (PE) versus delaying treatment with PE in altering neuroendocrine-related symptoms of post-traumatic stress disorder in women.

This single-blind study will randomly assign two thirds of participants to PE therapy immediately following a traumatic event and one third to a waitlist condition (WL), in which they will receive no treatment until a later date. Participants assigned to receive PE will do so once weekly for 10 weeks. Participants assigned to the WL condition will receive no treatment for 10 weeks, and then will begin PE therapy once weekly for an additional 10 weeks. Study visits will occur at baseline, Week 10, and 6 months post-treatment for those in both conditions, with additional visits 10 weeks and 6 months post-PE therapy for those in the WL condition. Psychological measurements to be assessed at these visits will include PTSD symptoms, anxiety, depression, and PTSD-related cognitions. Physical assessments will include urine and saliva tests, as well as a dexamethasone-suppression test. Participants in the PE condition will also provide saliva samples at points throughout the study to monitor changes in cortisol and catecholamines.

ELIGIBILITY:
Inclusion Criteria:

* Chronic post-traumatic stress disorder
* Minimum of 3 months passed since traumatic event happened
* Agree to use an effective form of contraception throughout the study

Exclusion Criteria:

* History of schizophrenia, bipolar disorder, or cognitive dysfunction due to a general medical condition
* History of alcohol or other drug abuse or dependence within 3 months of study enrollment
* Mental retardation or other pervasive developmental disorder
* Unwillingness or inability to discontinue current psychotherapy treatment (stable psychiatric medication therapy taken during the study is not criteria for exclusion)
* Significant risk of violence or history of serious violent behavior within one year of study enrollment
* Medically unstable condition
* Continuing intimate relationship with the perpetrator when the trauma involves assault
* At risk for suicide risk
* Currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2001-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
PTSD severity; measured by the PSS-I immediately after 10 weeks of treatment and at 6-month follow-up
Salivary cortisol; measured immediately after 10 weeks of treatment
Urinary cortisol and catecholamines; measured immediately after 10 weeks of treatment and at 6-month follow-up

SECONDARY OUTCOMES:
Depression; measured by the BDI immediately after 10 weeks of treatment and at 6-month follow-up
State-anxiety; measured by the STAI-S immediately after 10 weeks of treatment and at 6-month follow-up.
Trauma-related cognitions; measured by the PTCI immediately after 10 weeks of treatment and at 6-month follow-up
Salivary cortisol; measured at 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Edna B. Foa, Ph.D., Principal Investigator — University of Pennsylvania; Rachel Yehuda, Ph.D., Principal Investigator — Mt. Sinai School of Medicine
Locations (1):
- Center for the Treatment and Study of Anxiety, University of Pennsylvania, Philadelphia, Pennsylvania, United States